CLINICAL TRIAL: NCT02358460
Title: Randomised Controlled Trial Comparing Volume-targeted to Pressure-limited Ventilation in Infants Born at or Near Term
Brief Title: Pressure-limited Ventilation Versus Volume-targeted Ventilation in Term Newborns
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 07/H0808/147-3
Record Dates: First submitted 2015-01-13; First posted 2015-02-09 (Estimated); Last update posted 2015-02-09 (Estimated); Status verified 2015-02

CONDITIONS: Respiratory Insufficiency
Keywords: neonatal; respiratory; mechanical ventilation
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pressure-limited ventilation (Active Comparator)
  Interventions: Device: Ventilation delivered by SLE5000 ventilator
- Volume-targeted ventilation (Active Comparator)
  Interventions: Device: Ventilation delivered by SLE5000 ventilator

INTERVENTIONS:
Device: Ventilation delivered by SLE5000 ventilator — In pressure-limited ventilation arm, ventilator settings as required to maintain appropriate oxygenation and carbon-dioxide elimination.
  In volume-targeted ventilation arm, set target volume at 5ml/kg and wean rate. In both arms, aim to keep blood gases within normal limits.

SUMMARY:
A randomised controlled trial comparing volume-targeted ventilation to pressure-limited ventilation in infants born at or near term.

DETAILED DESCRIPTION:
Aims: There is increasing evidence that volume-targeted ventilation (VTV) holds benefits for preterm infants in comparison to pressure-limited ventilation. It is not known whether the same is true in the case of infants born at term. This study aims to compare pressure-limited to VTV in term-born infants.

Hypothesis: Volume-targeted will be associated with significantly earlier extubation compared to pressure-limited ventilation Primary outcome: Time to extubation. Methods: Ventilated infants 34 weeks or more gestational age at birth were recruited and randomly allocated to receive either pressure-limited or VTV. Adjustments to ventilator settings were made according to the trial protocol. Infants were deemed to have met failure criteria if they required HFOV or peak pressures of more than 30 cm of water. Analysis will be by intention-to-treat.

ELIGIBILITY:
Inclusion Criteria:

* Mechanically ventilated
* Born at gestation 34 weeks and above

Exclusion Criteria:

* Congenital diaphragmatic hernia
* Congenital heart disease

Ages: 1 Minute to 4 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2011-05; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Duration of mechanical ventilation | For each patient, the exact number of hours from the date and time of randomisation to the date and time of successful removal of the endotracheal tube, assessed up to 4 weeks.
  Data will be collected from the intensive care observation chart to determine the time at which the infant was successfully taken off of mechanical ventilation, assessed up to 4 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Greenough, MD, Principal Investigator — King's College Hospital NHS Trust
Locations (2):
- United Kingdom (2):
  - King's College Hospital NHS Foundation Trust, London, London
  - Neonatal Intensive Care Unit, London